CLINICAL TRIAL: NCT02361697
Title: Monitoring of Neurodegenerative Processes in Children With Multiple Sclerosis by Diffusion-weighed Magnetic Resonance Imaging (DTI)
Brief Title: DTI in Children With Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Muenster (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014-490-f-S
Record Dates: First submitted 2015-01-19; First posted 2015-02-12 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Multiple Sclerosis - Relapsing Remitting; Clinically Isolated Syndrome, CNS Demyelinating
Keywords: pediatric multiple sclerosis; clinically isolated syndrome in children; biomarker; magnetic resonance imaging; diffusion weighted imaging
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Demyelinating Diseases | interventions — Diffusion Tensor Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DTI-MRI (Other): MRI of the brain with specific DTI-sequences according to a specific investigation protocol
  Interventions: Other: DTI-MRI

INTERVENTIONS:
Other: DTI-MRI — MRI of the brain with special DTI-sequences are performed in each child with multiple sclerosis or clinically isolated syndrome at timepoint of first manifestation and every 6 months in a longterm follow-up of 3 years

SUMMARY:
This is a prospective, non-randomised, non-blinded, single center study of children and adolescents with multiple sclerosis and clinically isolated syndrome to detect differences or early changes in diffusion-weighted imaging (DTI) by magnetic resonance imaging (MRI).

DETAILED DESCRIPTION:
In children and adolescents with either multiple sclerosis or clinically isolated syndrome an MRI with special DTI-sequences of the brain is performed at timepoint of first manifestation of disease and every 6 months at 3 Tesla MRI according to a specific investigation protocol.

Besides MRI-DTI several clinical data are recorded every 6 months:

1. expanded disability status scale (EDSS)
2. disease activity/ relapse rate
3. lesion load (number of T2-lesions)
4. brain atrophy
5. visual and somatosensoric evoked potentials (VEP, SSEP)
6. neuropsychological examination

Furthermore a complete neurological examination is done every 6 months and particular medication of each patient is recorded in a specific investigator form (case report form, CRF)

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* diagnosis of multiple sclerosis (MS) according to the McDonald criteria 2010 and the consensus recommendations of International Pediatric MS Study Group (IPMSSG) (Krupp et al 2013)
* diagnosis of CIS according to the consensus recommendation of IPMSSG (Krupp et al 2013)
* all types of medication/therapy

Exclusion Criteria:

* pregnancy
* claustrophobia
* allergic reaction of gadolinium (contrast medium)
* implantation of cardiac device
* implantation of neurostimulators
* implantation of cochlea implants
* presence of tattooing (over 20% of body surface)
* presence of permanent-make-up
* presence of permanent transdermal patches
* presence of special catheter systems with temperature probes which cannot be removed
* implantation of metalliferous implants or implants which could contain metal traces
* implantation of artificial heart valves
* implantation of stents or coils
* presence of metal fragments in the eyes

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
change from baseline fractional anisotropy (FA) at 36 months measured by cerebral MRI and special DTI sequences | every 6 months (from date of randomization until the end of the study, assessed up to 36 months)
  measured by cerebral MRI and special DTI sequences
change from baseline apparent diffusion coefficient (ADC) at 36 months measured by cerebral MRI and special DTI sequences | every 6 months (from date of randomization until the end of the study, assessed up to 36 months)
  measured by cerebral MRI and special DTI sequences

SECONDARY OUTCOMES:
Disease activity (relapse rate, lesion load) | every 6 months (from date of randomization until the end of the study after 36 months)
  relapse rate, lesion load
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | every 6 months (from date of randomization until the end of the study, assessed up to 36 months)
EDSS (Expanded disability status scale, Values between 0-10) | every six months (from date of randomization until the end of the study, assessed up to 36 months)
  Expanded disability status scale, Values between 0-10
spinal lesion load measured by spinal MRI (which is performed in each participant every 12 months) | every 12 months (from date of randomization until the end of the study, assessed up to 36 months)
  measured by spinal MRI (which is performed in each participant every 12 months)
VEP-Score | every 6 months (from date of randomization until the end of the study, assessed up to 36 months)
  score of visual evoked potential (amplitudes, latency) Values between 0-4
SSEP somatosensory evoked potentials, records of amplitudes and latency | every 12 months (from date of randomization until the end of the study, assessed up to 36 months)
  somatosensory evoked potentials, records of amplitudes and latency
Medication particular medication of each patient | every 6 months (from date of randomization until the end of the study, assessed up to 36 months)
  particular medication of each patient
neurocognitive deficits neuropsychological test battery | every 12 months (from date of randomization until the end of the study, assessed up to 36 months)
  neuropsychological test battery including the following tests
  1. Standard Progressive Matrices (SPM)
  2. VLMT - verbal comprehension and retentivity test by Helmstaedter
  3. ROF - Rey-Osterrieth-Figure
  4. TMT A/B - Trail-Making-Test Form A and B
  5. RWT - Regensburg word fluency test
  6. block-span Corsi
  7. count span test
  8. SDMT - Symbol Digit Modalities Test
  9. BDI-II, Revision - Beck Depressions-Inventory
  10. PedsQL - Pediatric Quality of Life Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Christiane Elpers, MD, Principal Investigator — University Hospital Muenster
Locations (1):
- University Hospital Muenster, Münster, Germany